CLINICAL TRIAL: NCT06505148
Title: Comparing the Difference in Pain Control in the Pediatric General Surgery Population: to Alternate or Combine Acetaminophen and Ibuprofen?
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Baylor Scott and White Health (Other)
Responsible Party: Principal Investigator, Marlene Porter, Principal Investigator, Baylor Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 024-301
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Pediatric Disorder
Keywords: non opioid; pain management; pediatric pain; pediatric pain management
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: One group will be prescribed the acetaminophen and ibuprofen alternating every 3 hours. And the other group will be prescribed acetaminophen and ibuprofen combine treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will prescribe study participants in group 1 acetaminophen and ibuprofen alternating treatment every three hours. The dosage will be weight-based.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen
- Group B (Active Comparator): Group B will be prescribed acetaminophen and ibuprofen combined treatment every 6 hours. The dosage will be weight-based.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — administered alternatively with other drug
Drug: Ibuprofen — administered alternatively with other drug

SUMMARY:
To examine the difference in pain control in the pediatric general surgery population alternating acetaminophen and Ibuprofen q 3 hours vs giving them simultaneous combination therapy around the clock.

DETAILED DESCRIPTION:
The purpose of the study is to compare the difference in pain control in the pediatric general surgery population of those who receive alternating acetaminophen and ibuprofen every 3 hours to those who receive acetaminophen and ibuprofen combined therapy around the clock. Additionally, to investigate the difference in parent adherence to pain treatment plans between the alternating group from the combined group.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 3 years to 18 years
* General surgery service (hernia, appendectomy, chole, circumcision, wounds, vacs, implanted central line, etc.)

Exclusion Criteria:

* Patients who are allergic to acetaminophen and/or ibuprofen
* Patients being evaluated by SANE or evaluated for nonaccidental trauma
* Patients admitted post-op

The study will take place at McLane Children's Hospital Temple Market. Patients who are pregnant.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Faces, Legs, Activity, Cry, and Consolability (FLACC) pain assessment scale. | 24, 48, and 72 hours after surgery
  Pain will be assessed using an age-appropriate pain rating scale. The FLACC is an interval scale quantifying pain behavior with scores ranging from 0 no pain behaviors to 10 most possible pain behaviors. The five categories of behaviors assessed with the FLAC include facial expressions, leg movement, activity, crying, and consolability.
Pain Visual Analog Scale (VAS) | 24, 48, and 72 hours after surgery
  This tool portrays a 10cm ruler visual and the patient selects the marker indicating their pain intensity, 0 indicating no pain to 10 indicating the worst pain possible.
Numeric Pain Rating Scale (NPRS) | 24, 48, and 72 hours after surgery
  The NPRS is scored on an 11-point scale where the higher the number indicating severe more the pain.

SECONDARY OUTCOMES:
Parent/ guardian adherence | 72 hours after surgery
  Adherence will be assessed by asking the parent/guardian regarding their ability to follow pain regimen and the ease to follow the instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Health Temple Market, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data-sharing considerations will be addressed upon receipt of a formal request. Upon receipt of a formal request, data sharing will proceed once a data-sharing agreement has been established. The rationale for the data sharing plan is that data obtained for the study is considered proprietary to BSWH.